CLINICAL TRIAL: NCT03581084
Title: Inpatient Clinical Trial of NAC
Acronym: ICON
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was redesigned to be conducted in an outpatient setting.
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-24231; P01HL128191 (NIH)
Record Dates: First submitted 2018-04-12; First posted 2018-07-10 (Actual); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: This is a single-arm study which means all study participants will receive the same treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- N-acetylcysteine (Experimental): This study will look at the effects of a medication, called n-acetylcysteine or NAC, on lung function. NAC is already approved for use in people with chronic airway conditions, including asthma. However, it is not known who this medication works best in. We believe this medication will likely have the most benefit in people with asthma that have mucus in their airways or "mucus plugging." Initial study procedures will include lung function measurements, a low dose CT scan, a blood draw, and a sputum induction. The CT lung imaging will identify asthmatics with mucus plugs.
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — Research participants that meet the study inclusion criteria will be admitted to a medical-surgical ward in Moffitt-Long Hospital (UCSF Medical Center) for 6 days and 5 nights and treated with an inhaled mixture of NAC and albuterol four times per day spaced at 4 to 6 hours apart.

SUMMARY:
The purpose of this study is to determine the beneficial effect of n-acetylcysteine (NAC), an inhaled medication that breaks down mucus, on lung function. NAC is a medication approved by the US Food and Drug Administration (FDA) for the treatment of chronic diseases of the respiratory system, including asthma. With CT lung imaging, the investigators seek to identify a subgroup of patients with asthma with a 'mucus' profile. This is a single-arm study which means all participants will receive the same treatment.

DETAILED DESCRIPTION:
N-acetylcystine (NAC) is a mucolytic medication, meaning that it breaks apart mucus. Investigators know that mucus is a factor in severe asthma attacks. However, mucus may be a factor in chronic severe asthma as well. This role has been hard to prove because of difficulty in showing that mucus occludes the lumen in chronic severe disease. Using a novel approach of scoring mucus occlusion, investigators have used CT imaging to uncover that a majority of people with severe asthma have at least one lung segment with a mucus plug and 27% have more than four lung segments with mucus plugs.

Historically, studies of mucolytics, like NAC, have not shown benefit in other obstructive lung diseases, like COPD. However, utilizing CT mucus scores as a biomarker, investigators believe that mucolytic treatment may prove useful for those with significant mucus impaction.

This is a single-arm study of participants with asthma who also have evidence of mucus in their lungs as determined by CT imaging. Investigators hypothesize that by treating asthmatics, chosen based on the presence of mucus in the airways, with a mucolytic like NAC, will result in an improvement of lung function.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 80 years of age at Visit 1
2. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
3. Able to perform reproducible spirometry according to ATS criteria
4. Physiological evidence of airflow obstruction (FEV1 bronchodilator reversibility of ≥ 12% or hyperreactivity to methacholine reflected by a methacholine PC20 ≤ 16 mg/mL)
5. Clinical history of asthma per patient report or medical record
6. Pre-bronchodilator FEV1 > 35% predicted
7. Post-bronchodilator FEV1 > 40% but < 90% predicted
8. Asthma requiring treatment with inhaled corticosteroids (ICS) for 3 months or greater
9. CT mucus score > 3

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
3. Smoking of tobacco or other recreational inhalants in last year and/or >10 pack-year smoking history
4. Current participation in an investigational drug trial
5. Other chronic pulmonary disorders, including (but not limited to) cystic fibrosis, chronic obstructive pulmonary disease, chronic bronchitis, vocal cord dysfunction (that is the sole cause of respiratory symptoms and at the PI's discretion), severe scoliosis or chest wall deformities that affect lung function, or congenital disorders of the lungs or airways
6. Unwillingness to follow study procedures
7. History of allergy or intolerance to study drug
8. Any other criteria that places the subject at unnecessary risk according to the judgment of the Principal Investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fahy, M.D, M.Sc., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Hays SR, Fahy JV. The role of mucus in fatal asthma. Am J Med. 2003 Jul;115(1):68-9. doi: 10.1016/s0002-9343(03)00260-2. No abstract available. PMID 12867239
- [Background] DUNNILL MS. The pathology of asthma, with special reference to changes in the bronchial mucosa. J Clin Pathol. 1960 Jan;13(1):27-33. doi: 10.1136/jcp.13.1.27. PMID 13818688

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-acetylcysteine
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | N-acetylcysteine
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1
Forced Expiratory Volume in One Second (FEV1) Measurement [Number; unit: liters] | .85
Mean Number of Mucus Plugs [Mean (Full Range); unit: number of mucus plugs] — Number of mucus plugs identified by the radiologist on the chest CT scan. Independently reviewed by two radiologists, and the average number of mucus plugs is reported.
  number of mucus plugs | 11 [6 to 16]

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Measurement
Description: Post-treatment FEV1 is reported. FEV1 is measured via spirometry.
Time Frame: end of the one week treatment period
Measure: Number; unit: liters
Arm/Group | N-acetylcysteine
Number analyzed (Participants) | 1
liters | 0.86

2. Secondary Outcome: Computed Tomography (CT) Scan Mucus Score
Description: Post-treatment CT mucus scores will be compared to pre-treatment CT mucus score
Time Frame: From the start of the one week treatment period to the three month follow-up
Population: The researchers were unable to obtain a post-treatment CT scan for the enrolled subject and therefore have nothing to report for this outcome measure.
Arm/Group | N-acetylcysteine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events will be monitored by the Clinical PIs (Drs. Fahy, Woodruff and Lazarus) in real-time. Safety and tolerability data will be summarized quarterly. Adverse events will be tabulated and will include the number of patients for whom the event occurred, the rate of occurrence, and the severity and relationship to study drug. All AEs will be reviewed quarterly.
Arm/Group | N-acetylcysteine
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (N=1)
Angina (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (N=1)
Headache (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT03581084/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT03581084/SAP_001.pdf